CLINICAL TRIAL: NCT06605404
Title: Molecular Residual Disease in Solid Tumors: A Prospective Study to Collect Clinical Data and Biospecimens to Support Discovery and Development of Cancer Biomarkers
Brief Title: Pan-tumor MRD Study
Status: Recruiting | Type: Observational
Sponsor: Paradigm Health (Industry)
Responsible Party: Sponsor
Other Study IDs: FH-PrwS-07-002
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Muscle Invasive Bladder Urothelial Carcinoma; Esophageal Cancer; Gastric and Gastroesophageal Junction (GEJ) Adenocarcinoma; Melanoma (Skin Cancer); NSCLC (Non-small Cell Lung Cancer); Pancreatic (Exocrine Only); Mix of Solid Tumors (MOST)
Keywords: observational; biospecimen; routine care
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma; Melanoma; Carcinoma, Non-Small-Cell Lung | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood and tissue samples
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (7):
- Muscle Invasive Urothelial Carcinoma of the Bladder (MIBC): Muscle Invasive Urothelial Carcinoma of the Bladder (MIBC)
  Interventions: Diagnostic Test: blood and tissue samples; Other: blood and tissue samples
- Esophageal: Esophageal cancer
  Interventions: Diagnostic Test: blood and tissue samples; Other: blood and tissue samples
- Gastric and Gastroesophageal Junction (GEJ): Gastric and Gastroesophageal Junction (GEJ)
  Interventions: Diagnostic Test: blood and tissue samples; Other: blood and tissue samples
- Melanoma: Melanoma
  Interventions: Diagnostic Test: blood and tissue samples; Other: blood and tissue samples
- Non-small cell lung (NSCLC): Non-small cell lung (NSCLC)
  Interventions: Diagnostic Test: blood and tissue samples; Other: blood and tissue samples
- Pancreatic (exocrine only): Pancreatic (exocrine only)
  Interventions: Diagnostic Test: blood and tissue samples; Other: blood and tissue samples
- Mix of Solid Tumors (MOST): Mix of Solid Tumors (MOST)
  Interventions: Diagnostic Test: blood and tissue samples; Other: blood and tissue samples

INTERVENTIONS:
Diagnostic Test: blood and tissue samples — routine standard of care
Other: blood and tissue samples — Routine standard of care

SUMMARY:
The purpose of this observational study is to collect clinical information, blood, and tumor tissue samples from participants diagnosed with stage I, stage II, or operable stage III cancer in select solid tumors. The information collected will be used to develop tests to better understand cancer, for example, to improve cancer detection and to assess the risk of cancer coming back.

Participants will receive routine standard of care from their doctor and their involvement is expected to last for approximately five and a half (5.5) years.

ELIGIBILITY:
Eligibility Criteria:

1. Age 18 years or older.
2. Confirmed histological or cytological diagnosis of a malignant solid tumor that is either specified in one of the pre-defined tumor cohorts or meets the enrollment criteria for the Mix of Solid Tumors (MOST) cohort (Table 1).
3. Eligible for curative intent therapy, with surgical resection of cancer planned.

   a. If surgical resection has occurred, enrollment should occur within 3 months of surgical resection and before initiation of adjuvant therapy.
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2.
5. No systemic therapy for current cancer diagnosis administered before enrollment.
6. Willing and able to comply with required study procedures, including blood sample collection and primary tumor tissue submission from diagnostic biopsy or surgical excision.
7. Has completed all therapy (including endocrine therapy) 3 or more years ago for any previous invasive solid organ malignancy (with exception of nonmelanoma skin cancers) or hematologic malignancy. Individuals with a prior history of noninvasive (in situ) carcinomas may participate if they have received definitive treatment (no washout period required).
8. No concurrent diagnosis of another invasive cancer, except for nonmelanoma skin cancers.
9. No prior allogeneic hematopoietic stem cell transplant.
10. Able and willing to provide informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization for the release of personal health information.

    Cohort Specific Criteria
11. Muscle-invasive urothelial carcinoma of the bladder and Melanoma Cohorts: Stage II or operable III cancer:
12. Esophageal, Gastric/GEJ, and NSCLC Cohorts: Stage I, II, or operable III cancer.
13. Pancreatic Cohort: Stage I, II or operable III cancer, exocrine only disease.
14. MOST cohort: Stage II or operable stage III solid tumor diagnosis that meets eligibility criteria and is not included in the other cohorts.

The following tumor types are excluded:

1. Central nervous system (CNS) malignancies
2. Colorectal cancer
3. Breast cancer
4. Squamous cell skin cancer
5. Basal cell carcinoma
6. Gastrointestinal stromal tumors (GIST)
7. Thyroid cancer
8. Uveal melanoma
9. Low or intermediate grade neuroendocrine tumors

   ■ Eligible tumor types: High-grade neuroendocrine tumors, including neuroendocrine carcinomas, Merkel cell carcinomas, and small cell lung cancer are permissible
10. Hematologic cancers including multiple myeloma or other plasma cell dyscrasias, Hodgkin's lymphoma, non-Hodgkin's lymphoma, acute or chronic leukemias including chronic lymphocytic leukemia / small lymphocytic leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender as defined at birth
Study Population: Study participants diagnosed with stage I, stage II, or operable stage III cancer in select solid tumors
Sampling Method: Non-Probability Sample
Enrollment: 1350 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2032-04 (Estimated)

PRIMARY OUTCOMES:
Blood and tissue biospecimen registry | Observation from enrollment to 5.5 years after enrollment
  To establish a blood and tissue biospecimen resource in participants with operable solid tumors, with clinical, lab, radiographic, and pathology annotation for the discovery, development, and validation of MRD assays.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Medical Oncology Associates of San Diego, San Diego, California
  - Taylor Cancer Research Center, Maumee, Ohio

IPD SHARING:
Plan to Share IPD: No